CLINICAL TRIAL: NCT05437718
Title: Application of Ultrasound-Guided Thoracic Paravertebral Block in Pulmonary Ablation Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Yuan Zhou, Principal Investigator, Affiliated Hospital of Nantong University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2021-K145
Record Dates: First submitted 2022-06-12; First posted 2022-06-29 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms | interventions — Ropivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Group NB (thoracic paravertebral block Group) (Other): Thoracic paravertebral block(TPVB) is performed 20 minutes before the ablation surgery began,30 mL of 0.375% ropivacaine was totally injected in T3-4 and T5-6 spinal segment（the block segment can be adjusted according to the tumor site) under the ultrasound guidance.
  Interventions: Other: Ropivacaine

INTERVENTIONS:
Other: Ropivacaine — Thoracic paravertebral block(TPVB) is performed on the patients who undergo the thermal ablation therapy.

SUMMARY:
Local thermal ablation therapy of tumor is a rapidly developing minimally invasive therapy for lung tumors in recent years. This study evaluated the efficacy of thoracic paravertebral block (TPVB) for anaesthesia during ablation surgery of lung tumor.

DETAILED DESCRIPTION:
Lung cancer is a serious threat to human health and life. Local thermal ablation therapy of tumor is the focus of domestic and overseas research in the past decade.Thoracic paravertebral nerve block (TPVB) is the technique of injecting local anaesthetic in the paravertebral space to anesthetizes the spinal nerve roots and sympathetic chain，which will produces ipsilateral and somatic blockade.The present study was designed to evaluate the analgesic effect and safety of TPVB in the ablation surgery of lung tumor.

After obtaining approval from the Hospital Ethics Committee and informed written consent from the patients,30 adult patients scheduled for Local thermal ablation therapy of lung tumours were recruited. Patients were excluded if they had a history of psychiatric illness, chronic pain, regular analgesic usage or there were contraindications to performing a TPVB, such as chest wall deformity, severe coagulopathy, local infection and allergy to local anaesthetic drugs. The study lasted a total of six months.

During the preoperative visit, all patients received the explanation of overall research approach.After entering the CT fluoroscopy room, peripheral veins and routine monitoring that included electrocardiography, pulse oximetry, and noninvasive arterial blood pressure were obtained in all patients.Thoracic paravertebral block was performed 20 minutes before the Local thermal ablation therapy began.The degree of pain was assessed using VAS score; at performing TPVB，the beginning of surgery， 6 and 24 hours after ablation surgery.Dezocine will be given as remedial analgesia.Following the operation, transferred the patients to the observation area where the vital signs were monitored for 30 min.Assessing and record the degree of patients and surgeons satisfaction for anesthetic management.

ELIGIBILITY:
Inclusion criteria

1. Patients diagnosed with lung cancer by imaging examination
2. Informed consent of the patient and study approval by the Medical Ethics Committee

Exclusion criteria

1. have a history of psychiatric illness, chronic pain, regular analgesic usage
2. have contraindications to performing a TPVB, such as chest wall deformity, severe coagulopathy, local infection
3. have allergy to local anaesthetic drugs

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2022-05-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
The degree of pain that patients feel who undergo ablation surgery is assessed by the visual analog scale (VAS). | During surgery
  All patients are instructed on the use of the visual analog scale (VAS) for pain assessment before surgery, then anesthetist evaluate the analgesic effect of TPVB for the ablation surgery with the VAS during surgery(0="no pain"and 10=the "worst pain").

CONTACTS AND LOCATIONS:
Overall Officials: Yuan Zhou, Doctor, Study Director — Affiliated Hospital of Nantong University
Locations (1):
- Affiliated Hospital of Nantong University, Nantong, Jiangsu, China